CLINICAL TRIAL: NCT01059630
Title: An Open-Label, Multicenter, Randomized, Phase III Study to Investigate the Efficacy and Safety of Bendamustine Compared With Bendamustine+RO5072759 (GA101) in Patients With Rituximab-Refractory, Indolent Non-Hodgkin's Lymphoma
Brief Title: A Study to Investigate the Efficacy and Safety of Bendamustine Compared With Bendamustine+Obinutuzumab (GA101) in Participants With Rituximab-Refractory, Indolent Non-Hodgkin's Lymphoma (GADOLIN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAO4753g; GO01297 (Other: Hoffmann-La Roche); 2009-015504-25 (EudraCT Number)
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Results first posted 2016-11-17 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: follicular; follicular lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular | interventions — obinutuzumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bendamustine Alone (Active Comparator): Participants will receive bendamustine 120 milligrams per meter square (mg/m^2) Intravenous (IV) infusion on Days 1 and 2 of each 28-day cycle for up to six cycles.
  Interventions: Drug: Bendamustine
- Obinutuzumab + Bendamustine (Experimental): Induction phase: Participants will receive bendamustine 90 mg/m^2 IV on Days 2 and 3 of Cycle 1 and on Days 1 and 2 of Cycles 2-6 (28-day cycles) for the first 10 participants and on Days 1 and 2 of each 28-day cycle for Cycles 1-6 for remaining participants. Participants will also receive obinutuzumab 1000 mg IV infusion on Days 1, 8, and 15 of Cycle 1; Day 1 of Cycles 2-6.
  Maintenance phase: Participants with complete response (CR), partial response (PR) or stable response (SD) then will receive obinutuzumab 1000 mg IV infusion every 2 months until disease progression or for up to 2 years (whichever occurs first).
  Interventions: Drug: Obinutuzumab; Drug: Bendamustine

INTERVENTIONS:
Drug: Obinutuzumab — IV infusion.
  Other Names: RO5072759; GA101
  Arms: Obinutuzumab + Bendamustine
Drug: Bendamustine — IV infusion.

SUMMARY:
This open-label, multicenter, randomized Phase III study will investigate the efficacy, safety, pharmacokinetics and pharmacoeconomics of obinutuzumab (RO5072759, GA101) combined with bendamustine followed by continued obinutuzumab treatment (maintenance monotherapy) compared with bendamustine alone treatment in participants with rituximab-refractory indolent Non-Hodgkin's lymphoma (iNHL). The end of study was defined to when safety follow-up for all patients had been completed (2 years' safety follow-up from last dose).

ELIGIBILITY:
Inclusion Criteria:

* History of histologically documented, B-lymphocyte antigen cluster of differentiation 20 plus (CD20+), iNHL
* Refractory to any previous regimen containing rituximab (defined by participants who did not respond or who progressed during or up to 6 months after treatment with rituximab or a rituximab-containing regimen)
* Previously treated with a maximum of four unique chemotherapy containing treatment regimens
* All participants must have at least one bi-dimensionally measurable lesion (greater than [>]1.5 centimeters (cm) in its largest dimension by computed tomography [CT] scan)

Exclusion Criteria:

* Prior use of any monoclonal antibody (other than anti-CD20) within 3 months prior to the start of Cycle 1, prior treatment with obinutuzumab was not allowed
* Chemotherapy or other investigational therapy within 28 days prior to the start of Cycle 1
* Prior treatment with bendamustine (within 2 years of the start of Cycle 1)
* Prior allogeneic stem cell transplant
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* History of sensitivity to mannitol
* Central nervous system lymphoma or prior diffuse large B-cell lymphoma (DLBCL), histological evidence of transformation to high grade or diffuse large B-cell lymphoma
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) or any major episode of infection requiring treatment with intravenous antibiotics or hospitalization within 4 weeks
* Participants with a history of confirmed progressive multifocal leukoencephalopathy (PML)
* Vaccination with a live vaccine a minimum of 28 days prior to randomization
* Recent major surgery (within 4 weeks), other than for diagnosis
* Presence of positive test results for Hepatitis B surface antigen (HBsAg); antibody to hepatitis B core antigen [anti-HBc]) with detectable viral load (positive hepatitis B virus [HBV] deoxyribo-nucleic acid [DNA]) or Hepatitis C
* Participants with chronic hepatitis B or seropositive occult (HBV) infection
* Participants with seronegative occult HBV infection or past HBV infection (defined as anti-HBc positive and HBV DNA negative) could be eligible if they were willing to be followed according to the protocol for HBV DNA testing
* Participants positive for Hepatitis C virus (HCV) antibody were eligible only if polymerase chain reaction(PCR) was negative for HCV Ribonucleic acid (RNA)
* Known history of human immunodeficiency virus (HIV) seropositive status
* Positive test results for human T-lymphotropic virus type I (HTLV 1) virus in endemic countries
* Women who are pregnant or lactating
* Fertile men or women of childbearing potential unless 1) surgically sterile or 2) using an adequate measure of contraception such as oral contraceptives, intrauterine device, or barrier method of contraception in conjunction with spermicidal jelly
* Ongoing corticosteroid use >30 milligrams per day (mg/day) prednisone or equivalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2010-04-30 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (121):
- United States (33):
  - Southern Cancer Center, PC, Mobile, Alabama
  - Dr. Donald W. Hill, MD, FACP, Casa Grande, Arizona
  - Highlands Oncology Group, Rogers, Arkansas
  - Kaiser Permanente - Bellflower, Bellflower, California
  - Bay Area Cancer Research Group, LLC, Pleasant Hill, California
  - Sharp Memorial Hospital, San Diego, California
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - Washington DC VA Med Center; Hematology, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Florida; Division of Hematology/Oncology, Gainesville, Florida
  - Md Anderson Cancer Center Orlando, Orlando, Florida
  - Rush Cancer Institute, Chicago, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Simmons Cancer Institute, Springfield, Illinois
  - University of Iowa, Iowa City, Iowa
  - Univ Louisville School of Med, Louisville, Kentucky
  - New England Cancer Specialists, Scarborough, Maine
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Capitol Comprehensive CA Care, Jefferson City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Hematology Oncology Assoc SJ, Mount Holly, New Jersey
  - San Juan Oncology, Farmington, New Mexico
  - The Mark H. Zangmeister Ctr; Mid Ohio Onc/Hem Inc., Columbus, Ohio
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Pacific Oncology, PC, Portland, Oregon
  - OHSU Ctr for Health & Healing, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Sanford Health System, Sioux Falls, South Dakota
  - South Texas Inst of Cancer, Corpus Christi, Texas
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Univ of Wisconsin Hosp & Clin, Madison, Wisconsin
- Austria (3):
  - Lkh-Univ. Klinikum Graz, Graz
  - Lkh Salzburg - Univ. Klinikum Salzburg; Iii. Medizinische Abt., Salzburg
  - Medizinische Universität Wien, Vienna
- Belgium (3):
  - ZNA Stuivenberg, Antwerp
  - AZ Groeninge, Kortrijk
  - CHU Ambroise Paré, Mons
- Canada (11):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Kelowna, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Manitoba Cancer Care, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Toronto East General Hospital; Main Pharmacy G Wing Basement, East York, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUM-Hosp Notre Dame, Montreal, Quebec
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
  - CHA Hopital de I enfant-Jesus, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Czechia (3):
  - Fakultni nemocnice Brno; Interni hematologicka a onkologicka klinika, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - I Interni klinika; Vseobecna fakultni nemocnice, Prague
- France (20):
  - Institut Bergonie; Hematologie Oncologie, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - Hopital Henri Mondor, Créteil
  - CH Dijon, Dijon
  - Centre d'oncologie-radiotherap, LeMans
  - Hopital Claude Huriez, Lille
  - Centre Leon Berard, Lyon
  - Hopital Bon Secour, Metz
  - CHU Hopital Saint Eloi, Montpellier
  - Hopital Hotel Dieu Et Hme; Clinique Dermatologique, Nantes
  - Hopital Necker, Paris
  - Hopital Saint Louis; Dermatologie 1, Paris
  - CHU Bordeaux, Pessac
  - Centre Hospitalier Lyon Sud; Hematolgie, Pierre-Bénite
  - Chu De Poitiers; Chu La Miletrie, Poitiers
  - CHU de Reims, Reims
  - Hopital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Clinique Ste Anne, Strasbourg
  - CHRU de; Maladies, Vasculaires, Vandœuvre-lès-Nancy
- Germany (6):
  - St. Johannes Hospital Duisburg, Duisburg
  - Klinikum Frankfurt Höchst, Frankfurt am Main
  - Asklepios Klinik St. Georg, Hamburg
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum der Universitat Munchen, Campus Grobhadern;; Medizinische Klinik und Poliklinik III, München
  - Schwarzwald-Baar Klinikum GmbH, Villingen-Schwenningen
- Italy (11):
  - Ospedale Vito Fazzi, Lecce, Apulia
  - Azienda Ospedaliera Universitaria di Modena, Modena, Emilia-Romagna
  - Azienda Ospedaliera Univ, Ematologica, Udine, Friuli Venezia Giulia
  - Azienda Ospedaliera Univ, Rome, Lazio
  - Universita La Sapienza, Rome, Lazio
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 2, Milan, Lombardy
  - Irccs Policlinico San Matteo; Divisione Di Ematologia, Pavia, Lombardy
  - Azienda Ospedale San Giovanni, Turin, Piedmont
  - Ospedale Mauriziano Umberto I, Turin, Piedmont
  - Azienda Ospedaliero Univ, Catania, Sicily
  - Azienda Ospedaliera Univ, Florence, Tuscany
- Netherlands (6):
  - VU MEDISCH CENTRUM; Dept. of Medical Oncology, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus Mc - Daniel Den Hoed Kliniek; Medical Oncology, Rotterdam
  - Erasmus MC, Rotterdam
  - Haga Ziekenhuis, The Hague
- Russia (8):
  - Regional Oncology Hospital, Irkutsk
  - Blokhin Cancer Research Center; Combined Treatment, Moscow
  - City Clin Hosp n.a. S.P.Botkin, Moscow
  - Russian Hema Res Ctr of RAMS, Moscow
  - Republican Clinical Hospital n.a. Baranov; Haematology, Petrozavodsk
  - Ryazan Regional Clinical Hosp, Ryazan
  - SRI of Hematology and Transfusiology, Saint Petersburg
  - St. Petersburg State Medical University n.a. I.P. Pavlov; Hematology, transfusiology and transplanta, Saint Petersburg
- Spain (5):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Univ. Nuestra Señora de Valme;, Sevillac, Sevilla
  - Hospital Universitario Basurto, Bilbao, Vizcaya
  - Hospital Universitario de la Princesa; Servicio de Hematologia, Madrid
  - Hospital Universitario La Paz, Madrid
- Sweden (4):
  - Skånes University Hospital, Skånes Department of Onclology, Lund
  - Hematology Center; Karolinska Univ Hosp, Stockholm
  - Norrlands Uni Hospital; Onkologi Avd., Umeå
  - Onc Clin, Akademiska Sjukhuset, Uppsala
- Switzerland (3):
  - Universitaetsspital Basel; Onkologie, Basel
  - Inselspital Bern; Universitätsklinik für medizinische Onkologie, Bern
  - Kantonsspital Graubünden;Onkologie und Hämatologie, Chur
- United Kingdom (5):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Leicester Royal Infirmary, Leicester
  - Barts & London School of Med; Medical Oncology, London
  - Freeman Hospital, Newcastle upon Tyne
  - Singleton Hospital; Pharmacy Department, Swansea

REFERENCES:
- [Derived] Pott C, Sehn LH, Belada D, Gribben J, Hoster E, Kahl B, Kehden B, Nicolas-Virelizier E, Spielewoy N, Fingerle-Rowson G, Harbron C, Mundt K, Wassner-Fritsch E, Cheson BD. MRD response in relapsed/refractory FL after obinutuzumab plus bendamustine or bendamustine alone in the GADOLIN trial. Leukemia. 2020 Feb;34(2):522-532. doi: 10.1038/s41375-019-0559-9. Epub 2019 Aug 28. PMID 31462735
- [Derived] Gibiansky E, Gibiansky L, Buchheit V, Frey N, Brewster M, Fingerle-Rowson G, Jamois C. Pharmacokinetics, exposure, efficacy and safety of obinutuzumab in rituximab-refractory follicular lymphoma patients in the GADOLIN phase III study. Br J Clin Pharmacol. 2019 Sep;85(9):1935-1945. doi: 10.1111/bcp.13974. Epub 2019 Jul 12. PMID 31050355
- [Derived] Cheson BD, Chua N, Mayer J, Dueck G, Trneny M, Bouabdallah K, Fowler N, Delwail V, Press O, Salles G, Gribben JG, Lennard A, Lugtenburg PJ, Fingerle-Rowson G, Mattiello F, Knapp A, Sehn LH. Overall Survival Benefit in Patients With Rituximab-Refractory Indolent Non-Hodgkin Lymphoma Who Received Obinutuzumab Plus Bendamustine Induction and Obinutuzumab Maintenance in the GADOLIN Study. J Clin Oncol. 2018 Aug 1;36(22):2259-2266. doi: 10.1200/JCO.2017.76.3656. Epub 2018 Mar 27. PMID 29584548
- [Derived] Sehn LH, Chua N, Mayer J, Dueck G, Trneny M, Bouabdallah K, Fowler N, Delwail V, Press O, Salles G, Gribben J, Lennard A, Lugtenburg PJ, Dimier N, Wassner-Fritsch E, Fingerle-Rowson G, Cheson BD. Obinutuzumab plus bendamustine versus bendamustine monotherapy in patients with rituximab-refractory indolent non-Hodgkin lymphoma (GADOLIN): a randomised, controlled, open-label, multicentre, phase 3 trial. Lancet Oncol. 2016 Aug;17(8):1081-1093. doi: 10.1016/S1470-2045(16)30097-3. Epub 2016 Jun 23. PMID 27345636

RESULTS

PARTICIPANT FLOW:
Groups:
- Bendamustine Alone: Participants received Bendamustine 120 mg/m^2 IV infusion on Days 1 and 2 of each 28-day cycle for up to six cycles.
- Obinutuzumab + Bendamustine: Induction phase: Participants received Bendamustine 90 mg/m^2 IV on Days 2 and 3 of Cycle 1 and on Days 1 and 2 of Cycles 2-6 (28-day cycles) for the first 10 participants and on Days 1 and 2 of each 28-day cycle for Cycles 1-6 for remaining participants. Participants also received obinutuzumab 1000 mg IV infusion on Days 1, 8, and 15 of Cycle 1; Day 1 of Cycles 2-6. Maintenance phase: Participants with CR, PR or SD then received obinutuzumab 1000 mg IV infusion every 2 months until disease progression or for up to 2 years (whichever occurred first).
Period: Overall Study
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Started | 209 | 204
Completed | 82 | 101
Not Completed | 127 | 103
Not completed — Death | 100 | 84
Not completed — Lost to Follow-up | 4 | 1
Not completed — Physician Decision | 2 | 4
Not completed — Withdrawal by Subject | 21 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine | Total
Number analyzed (Participants) | 209 | 204 | 413
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (11.5) | 62.0 (11.3) | 61.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 88 | 175
  Male | 122 | 116 | 238
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 174 | 183 | 357
  Not Stated | 30 | 15 | 45
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 3 | 6 | 9
  Black or African American | 3 | 5 | 8
  Multiple | 1 | 0 | 1
  Unknown | 19 | 12 | 31
  White | 181 | 180 | 361

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progressive Disease (PD) as Assessed by Independent Review Committee (IRC) or Death
Description: PD was assessed by an IRC according to the modified response criteria for indolent Non-Hodgkin's Lymphoma (iNHL) (Modified Cheson et al, 2007). PD was defined as appearance of any new lesion more than 1.5 centimeters (cm) in any axis during or at the end of therapy, even if other lesions are decreasing in size; at least a 50 percent (%) increase from nadir in the sum of product diameter (SPD) of any previously involved nodes, or in a single involved node, or the size of other lesions (example: splenic or hepatic nodules). To be considered PD, a lymph node with a diameter of the short axis of less than (<) 1.0 cm must increase by greater than or equal to (≥) 50% and to a size of 1.5 multiplied by 1.5 cm or more than 1.5 cm in the long axis; at least a 50% increase in the longest diameter of any single previously identified node greater than (>) 1 cm in its short axis.
Time Frame: Baseline until PD or death, whichever occurred first (assessed at baseline, 14 days prior to Cycle [Cy] 4 Day 1 [1 Cy=28days], 28-42 days after Cy 6 Day 1, then every 3 months up to 2 years and every 6 months for next 2 years [up to 4.5 years overall])
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
participants | 125 | 87

2. Primary Outcome: Progression-Free Survival (PFS) as Assessed by IRC
Description: PFS was defined as the time from randomization to the first occurrence of PD or death as assessed by an IRC according to the modified response criteria for iNHL (Modified Cheson et al, 2007). PD was defined as appearance of any new lesion more than 1.5 cm in any axis during or at the end of therapy, even if other lesions are decreasing in size; at least a 50% increase from nadir in the SPD of any previously involved nodes, or in a single involved node, or the size of other lesions (e.g., splenic or hepatic nodules). To be PD, a lymph node with a diameter of the short axis of <1.0 cm must increase by ≥ 50% and to a size of 1.5 multiplied by 1.5 cm or more than 1.5 cm in the long axis; at least a 50% increase in the longest diameter of any single previously identified node >1 cm in its short axis. PFS was estimated using Kaplan-Meier method and 95% confidence interval (CI) for median was computed using the method of Brookmeyer and Crowley.
Time Frame: Baseline until PD or death, whichever occurred first (assessed at baseline, 14 days prior to Cy 4 Day 1 [1 Cy=28days], 28-42 days after Cy 6 Day 1, then every 3 months up to 2 years and every 6 months for next 2 years [up to 4.5 years overall])
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
months | 14.1 [11.7 to 16.6] | 29.2 [20.5 to NA] — Upper limit was not reached due to low number of participants with events.
Statistical Analysis 1: Comparison: Bendamustine Alone vs Obinutuzumab + Bendamustine; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.40 to 0.70]

3. Secondary Outcome: Number of Participants With PD or Death as Assessed by Investigator
Description: PD was assessed by an investigator according to the modified response criteria for iNHL (Modified Cheson et al, 2007). PD was defined as appearance of any new lesion more than 1.5 cm in any axis during or at the end of therapy, even if other lesions are decreasing in size; at least a 50% increase from nadir in the SPD of any previously involved nodes, or in a single involved node, or the size of other lesions (e.g., splenic or hepatic nodules). To be considered PD, a lymph node with a diameter of the short axis of <1.0 cm must increase by ≥ 50% and to a size of 1.5 multiplied by 1.5 cm or more than 1.5 cm in the long axis; at least a 50% increase in the longest diameter of any single previously identified node >1 cm in its short axis.
Time Frame: Baseline until PD or death, whichever occurred first (up to 8.5 years overall))
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
participants | 152 | 132

4. Secondary Outcome: PFS as Assessed by Investigator
Description: PFS was defined as the time from randomization to the first occurrence of PD as assessed by an investigator according to the modified response criteria for iNHL (Modified Cheson et al, 2007), or death from any cause on study. PD was defined as appearance of any new lesion more than 1.5 cm in any axis during or at the end of therapy, even if other lesions are decreasing in size; at least a 50% increase from nadir in the SPD of any previously involved nodes, or in a single involved node, or the size of other lesions (e.g., splenic or hepatic nodules). To be considered PD, a lymph node with a diameter of the short axis of <1.0 cm must increase by ≥ 50% and to a size of 1.5 multiplied by 1.5 cm or more than 1.5 cm in the long axis; at least a 50% increase in the longest diameter of any single previously identified node >1 cm in its short axis. PFS was estimated using Kaplan-Meier method and 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: Baseline until PD or death, whichever occurred first (up to 8.5 years overall)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
months | 14.1 [12.6 to 16.2] | 25.8 [20.1 to 36.5]
Statistical Analysis 1: Comparison: Bendamustine Alone vs Obinutuzumab + Bendamustine; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.45 to 0.73]

5. Secondary Outcome: Percentage of Participants With Objective Response as Assessed by IRC
Description: Objective response was defined as having CR or PR as assessed according to the modified response criteria for iNHL (Modified Cheson et al, 2007). CR: Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present prior to therapy, liver and spleen have returned to normal size (if enlarged at baseline), If the bone marrow was involved by lymphoma prior to treatment, the infiltrate must have cleared on repeat bone marrow biopsy. PR: at least 50% regression of measurable disease compared to tumors measured by a baseline scan and no new sites; no increase in the size of the other nodes, liver, or spleen; with the exception of splenic and hepatic nodules, involvement of other organs is usually assessable and no measurable disease should be present. IRC review was performed up clinical cutoff date of to 1 May 2015.
Time Frame: Baseline until PD or death, whichever occurred first (up to approximately 5 years)
Population: ITT population. Here, number of participants analyzed signified those participants who had at least one post-baseline assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
percentage of participants | 77.5 [71.24 to 82.98] | 75.5 [69.00 to 81.23]
Statistical Analysis 1: Comparison: Bendamustine Alone vs Obinutuzumab + Bendamustine; Test type: Superiority or Other; p = 0.9298, Cochran-Mantel-Haenszel; Difference in response rate = 0.98, 95% CI 2-sided [0.58 to 1.65]

6. Secondary Outcome: Percentage of Participants With Objective Response as Assessed by Investigator
Description: Objective response was defined as having CR or PR as assessed according to the modified response criteria for iNHL (Modified Cheson et al, 2007). CR: Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present prior to therapy, liver and spleen have returned to normal size (if enlarged at baseline), If the bone marrow was involved by lymphoma prior to treatment, the infiltrate must have cleared on repeat bone marrow biopsy. PR: at least 50% regression of measurable disease compared to tumors measured by a baseline scan and no new sites; no increase in the size of the other nodes, liver, or spleen; with the exception of splenic and hepatic nodules, involvement of other organs is usually assessable and no measurable disease should be present.
Time Frame: Baseline until PD or death, whichever occurred first (up to approximately 8.5 years)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
percentage of participants | 83.3 [77.49 to 88.05] | 82.4 [76.42 to 87.32]
Statistical Analysis 1: Comparison: Bendamustine Alone vs Obinutuzumab + Bendamustine; Test type: Superiority or Other; p = 0.7857, Cochran-Mantel-Haenszel; Difference in response rate = -0.90, 95% CI 2-sided [-8.44 to 6.64]

7. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) as Assessed by IRC
Description: BOR observed during assessment period according to modified response criteria for iNHL (Modified Cheson et al, 2007). CR: complete disappearance of all detectable clinical evidence of disease & disease-related symptoms if present prior to therapy, PR: at least 50% regression of measurable disease compared to tumors measured by baseline scan & no new sites; no increase in size of other nodes, liver, or spleen; with exception of splenic & hepatic nodules, involvement of other organs is usually assessable & no measurable disease should be present, SD: Failing to attain criteria needed for a CR/PR, but not fulfilling those for PD, PD: appearance of any new lesion >1.5 cm in any axis during or at end of therapy, even if other lesions are decreasing in size; at least a 50% increase from nadir in SPD of any previously involved nodes, or in single involved node, or size of other lesions (e.g., splenic or hepatic nodules). IRC review was performed up clinical cutoff date of to 1 May 2015.
Time Frame: Baseline until PD or death, whichever occurred first (up to approximately 5 years)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
percentage of participants
  CR | 17.2 [12.37 to 23.04] | 16.2 [11.40 to 21.96]
  PR | 60.3 [53.31 to 66.97] | 59.3 [52.23 to 66.12]
  SD | 12.0 [7.89 to 17.15] | 13.7 [9.32 to 19.22]
  PD | 5.7 [3.00 to 9.81] | 4.9 [2.38 to 8.83]
  Unable to evaluate | 1.0 [0.12 to 3.41] | 1.0 [0.12 to 3.50]
  Missing | 3.8 [1.67 to 7.40] | 4.9 [2.38 to 8.83]

8. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) as Assessed by Investigator
Description: BOR: best response for a participant, observed during assessment period according to modified response criteria for iNHL (Modified Cheson et al, 2007). CR: complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present prior to therapy, PR: at least 50% regression of measurable disease compared to tumors measured by baseline scan and no new sites; no increase in size of other nodes, liver, or spleen; with exception of splenic and hepatic nodules, involvement of other organs is usually assessable and no measurable disease should be present, SD: Failing to attain the criteria needed for a CR or PR, but not fulfilling those for PD, PD: appearance of any new lesion more than 1.5 cm in any axis during or at the end of therapy, even if other lesions are decreasing in size; at least a 50% increase from nadir in the SPD of any previously involved nodes, or in single involved node, or the size of other lesions (e.g., splenic or hepatic nodules).
Time Frame: Baseline until PD or death, whichever occurred first (up to approximately 8.5 years)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
percentage of participants
  CR | 21.5 [16.16 to 27.73] | 23.5 [17.89 to 29.96]
  PR | 61.7 [54.76 to 68.34] | 58.8 [51.74 to 65.65]
  SD | 6.7 [3.71 to 10.98] | 6.4 [3.44 to 10.65]
  PD | 4.8 [2.32 to 8.62] | 6.4 [3.44 to 10.65]
  Unable to evaluate | 1.4 [0.30 to 4.14] | 0.5 [0.01 to 2.70]
  Missing | 3.8 [1.67 to 7.40] | 4.4 [2.04 to 8.21]

9. Secondary Outcome: Percentage of Participants With BOR at the End of Induction Treatment as Assessed by IRC
Description: BOR observed during assessment period according to modified response criteria for iNHL (Modified Cheson et al, 2007). CR: complete disappearance of all detectable clinical evidence of disease & disease-related symptoms if present prior to therapy, PR: at least 50% regression of measurable disease compared to tumors measured by a baseline scan & no new sites; no increase in size of other nodes, liver or spleen; with exception of splenic & hepatic nodules, involvement of other organs is usually assessable & no measurable disease should be present, SD: Failing to attain criteria needed for a CR/PR, but not fulfilling those for PD, PD: appearance of any new lesion >1.5 cm in any axis during or at end of therapy, even if other lesions are decreasing in size; at least a 50% increase from nadir in the SPD of any previously involved nodes, or in a single involved node, or size of other lesions (e.g., splenic/hepatic nodules). IRC review was performed up clinical cutoff date of to 1 May 2015.
Time Frame: Baseline until end of induction treatment (assessed at baseline, 14 days prior to Cy 4 Day 1 [1 Cy=28days], 28-42 days after Cy 6 Day 1)
Population: ITT population. Here, number of participants analyzed signified those participants who had reached the end of induction treatment response assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
percentage of participants
  CR | 12.0 [7.93 to 17.23] | 11.8 [7.69 to 17.00]
  PR | 52.4 [45.38 to 59.35] | 54.9 [47.80 to 61.86]
  SD | 10.1 [6.36 to 15.02] | 11.8 [7.69 to 17.00]
  PD | 10.6 [6.75 to 15.58] | 8.8 [5.31 to 13.59]
  Unable to Evaluate | 2.9 [1.07 to 6.17] | 2.0 [0.54 to 4.94]
  Missing | 12.0 [7.93 to 17.23] | 10.8 [6.88 to 15.87]

10. Secondary Outcome: Percentage of Participants With BOR at the End of Induction Treatment as Assessed by Investigator
Description: BOR: best response for a participant, observed during assessment period according to modified response criteria for iNHL (Modified Cheson et al, 2007). CR: complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present prior to therapy, PR: at least 50% regression of measurable disease compared to tumors measured by a baseline scan and no new sites; no increase in size of other nodes, liver, or spleen; with exception of splenic and hepatic nodules, involvement of other organs is usually assessable and no measurable disease should be present, SD: Failing to attain criteria needed for a CR or PR, but not fulfilling those for PD, PD: appearance of any new lesion more than 1.5 cm in any axis during or at the end of therapy, even if other lesions are decreasing in size; at least a 50% increase from nadir in the SPD of any previously involved nodes, or in a single involved node, or the size of other lesions (e.g., splenic or hepatic nodules).
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
percentage of participants
  CR | 15.8 [11.12 to 21.45] | 17.2 [12.25 to 23.04]
  PR | 53.1 [46.10 to 60.03] | 60.3 [53.23 to 67.06]
  SD | 4.3 [1.99 to 8.02] | 3.9 [1.71 to 7.58]
  PD | 12.0 [7.89 to 17.15] | 9.3 [5.70 to 14.16]
  Unable to Evaluate | 2.9 [1.06 to 6.14] | 0.5 [0.01 to 2.70]
  Missing | 12.0 [7.89 to 17.15] | 8.8 [5.31 to 13.59]

11. Secondary Outcome: Percentage of Participants With Objective Response at the End of Induction Treatment as Assessed by IRC
Description: as for outcome 5
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
percentage of participants | 64.4 [57.51 to 70.92] | 66.7 [59.75 to 73.10]
Statistical Analysis 1: Comparison: Bendamustine Alone vs Obinutuzumab + Bendamustine; Test type: Superiority or Other; p = 0.8347, Cochran-Mantel-Haenszel; Difference in response rate = 2.24, 95% CI 2-sided [-7.20 to 11.69]

12. Secondary Outcome: Percentage of Participants With Objective Response at the End of Induction Treatment as Assessed by Investigator
Description: as for outcome 6
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
percentage of participants | 68.9 [62.15 to 75.11] | 77.5 [71.09 to 82.99]
Statistical Analysis 1: Comparison: Bendamustine Alone vs Obinutuzumab + Bendamustine; Test type: Superiority or Other; p = 0.0466, Cochran-Mantel-Haenszel; Difference in response rate = 8.55, 95% CI 2-sided [-0.22 to 17.32]

13. Secondary Outcome: Duration of Response (DoR) as Assessed by IRC
Description: DoR: time from first objective response of CR/PR to first occurrence of PD/relapse/death from any cause. CR: Complete disappearance of all detectable evidence of disease & disease-related symptoms if present before therapy; liver, spleen returned to normal size; if bone marrow involved by lymphoma before treatment, infiltrate must be cleared on repeat bone marrow biopsy. PR: at least 50% measurable disease regressed vs. to baseline scan and no new sites; no increase in size of other nodes/liver/spleen, exception: splenic, hepatic nodules; other organs involved is usually assessable; no measurable disease present. PD: any new lesion >1.5 cm in any axis appear during or at end of therapy, even if other lesions are decreasing in size; at least 50% increase from nadir in SPD of any previously involved nodes, or in single involved node, or size of other lesions. DoR estimated using Kaplan-Meier method. IRC review performed up to clinical cutoff date 1 May 2015.
Time Frame: Baseline until PD or death, whichever occurred first (up to approximately 5 years)
Population: ITT population. Here, number of participants analyzed signified those participants who had objective response at any time during the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 165 | 158
months | 12.7 [10.4 to 14.1] | 38.5 [25.4 to NA] — Upper limit of 95% confidence interval could not be reached due to low number of participants with events.
Statistical Analysis 1: Comparison: Bendamustine Alone vs Obinutuzumab + Bendamustine; Test type: Superiority or Other; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.31 to 0.61]

14. Secondary Outcome: Duration of Response (DoR) as Assessed by Investigator
Description: DoR: time from first objective response of CR/PR to first occurrence of PD/relapse/death from any cause. CR: Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present prior to therapy; liver, spleen returned to normal size (if enlarged at baseline); if bone marrow was involved by lymphoma prior to treatment, infiltrate must have cleared on repeat bone marrow biopsy. PR: at least 50% regression of measurable disease compared to baseline scan and no new sites; no increase in size of other nodes, liver, or spleen; with exception of splenic, hepatic nodules; involvement of other organs is usually assessable; no presence of measurable disease. PD: appearance of any new lesion >1.5 cm in any axis during or at end of therapy, even if other lesions are decreasing in size; at least 50% increase from nadir in SPD of any previously involved nodes, or in single involved node, or size of other lesions. DoR was estimated using Kaplan-Meier method.
Time Frame: Baseline until PD or death, whichever occurred first (up to approximately 8.5 years)
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
months | 12.7 [11.1 to 15.5] | 32.3 [20.8 to 39.0]
Statistical Analysis 1: Comparison: Bendamustine Alone vs Obinutuzumab + Bendamustine; Test type: Superiority or Other; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.39 to 0.67]

15. Secondary Outcome: Disease-Free Survival (DFS) in Participants With CR as Assessed by IRC
Description: DFS was defined as the time from the first occurrence of a documented CR until progression on the basis of the IRC assessments (as per modified response criteria for iNHL [Modified Cheson et al, 2007]) or death from any cause on study. CR: Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present prior to therapy, liver and spleen have returned to normal size (if enlarged at baseline), If the bone marrow was involved by lymphoma prior to treatment, the infiltrate must have cleared on repeat bone marrow biopsy. PD: appearance of any new lesion >1.5 cm in any axis during or at end of therapy, even if other lesions are decreasing in size; at least a 50% increase from nadir in SPD of any previously involved nodes, or in a single involved node, or size of other lesions. DFS was estimated using Kaplan-Meier method. IRC review was performed up clinical cutoff date of to 1 May 2015.
Time Frame: Baseline until PD or death, whichever occurred first (up to approximately 5 years)
Population: ITT population. Here, number of participants analyzed signified those participants who had an objective response of CR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 37 | 46
months | 13.2 [8.5 to NA] — Upper limit of 95% confidence interval could not be estimated due to low number of participants with events. | NA [NA to NA] — Median and 95% confidence interval could not be estimated due to low number of participants with events.
Statistical Analysis 1: Comparison: Bendamustine Alone vs Obinutuzumab + Bendamustine; Test type: Superiority or Other; Hazard Ratio (HR) = 0.13, 95% CI 2-sided [0.04 to 0.45]

16. Secondary Outcome: Disease-Free Survival (DFS) in Participants With CR as Assessed by Investigator
Description: DFS was defined as the time from the first occurrence of a documented CR until progression on the basis of the IRC assessments (as per modified response criteria for iNHL [Modified Cheson et al, 2007]) or death from any cause on study. CR: Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present prior to therapy, liver and spleen have returned to normal size (if enlarged at baseline), If the bone marrow was involved by lymphoma prior to treatment, the infiltrate must have cleared on repeat bone marrow biopsy. PD: appearance of any new lesion >1.5 cm in any axis during or at end of therapy, even if other lesions are decreasing in size; at least a 50% increase from nadir in SPD of any previously involved nodes, or in a single involved node, or size of other lesions. DFS was estimated using Kaplan-Meier method.
Time Frame: Baseline until PD or death, whichever occurred first (up to approximately 8.5 years)
Population: ITT population. Here, number of participants analyzed signified those participants who had an objective response of CR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
months | 20.0 [8.6 to 31.0] | 36.0 [26.6 to 68.2]
Statistical Analysis 1: Comparison: Bendamustine Alone vs Obinutuzumab + Bendamustine; Test type: Superiority or Other; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.29 to 0.81]

17. Secondary Outcome: Event-free Survival (EFS) as Assessed by IRC
Description: EFS was defined as the time between the date of randomization and the date of PD/relapse based on IRC assessments (as per modified response criteria for iNHL [Modified Cheson et al, 2007]), death from any cause on study, or start of a new anti-lymphoma therapy. PD: appearance of any new lesion >1.5 cm in any axis during or at end of therapy, even if other lesions are decreasing in size; at least a 50% increase from nadir in SPD of any previously involved nodes, or in a single involved node, or size of other lesions. EFS was estimated using Kaplan-Meier method. IRC review was performed up clinical cutoff date of to 1 May 2015.
Time Frame: Baseline until PD or death, whichever occurred first (up to approximately 5 years)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
months | 13.7 [11.4 to 15.5] | 25.3 [13.9 to 35.0]
Statistical Analysis 1: Comparison: Bendamustine Alone vs Obinutuzumab + Bendamustine; Test type: Superiority or Other; p = 0.0001, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.44 to 0.74]

18. Secondary Outcome: Percentage of Participants Who Died
Time Frame: Baseline until death (up to 8.5 years overall)
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 203 | 204
percentage of participants | 49.3 | 41.2

19. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time between the date of randomization and the date of death from any cause. OS was estimated using Kaplan-Meier method and 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: Baseline until death (up to 8.5 years overall)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
months | 65.6 [48.5 to 87.8] | 88.3 [71.1 to NA] — Data could not be estimated due to higher (>50%) number of censored participants.
Statistical Analysis 1: Comparison: Bendamustine Alone vs Obinutuzumab + Bendamustine; Test type: Superiority or Other; p = 0.0810, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.57 to 1.03]

20. Secondary Outcome: Change From Baseline (CFB) in Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym)-Physical Well Being Sub-scale Score
Description: The FACT-Lym measures 5 sub-scales which includes 42 items; responses to each item range from 0, "Not at all" to 4, "Very much". Total score ranges from 0-168. Physical Well-being sub-scale includes 7 items measured on 0-4 point scale. The total score for physical well-being sub-scale is sum of each 7 items (range: 0-28). Higher scores indicate a better participant-reported outcome (PRO)/quality of life (QoL). In timeframe, follow-up months represents months after end of induction (e.g. Follow-up Month 2 is 2 months after end of induction) and extension follow-up months represents months after end of 2 years normal follow-up (e.g. extension follow-up Month 6 is 6 months after end of normal 2 year follow-up).
Time Frame: Baseline, Day 1 of Cycles 3, 4, 5, End of induction treatment (up to Month 6); Follow-up Months 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, Final Follow-up (up to 2 years after end of induction); Extension follow-up Months 6, 18 and 24
Population: ITT population. Here, number of participants analyzed signified those participants who were evaluable for this outcome and "n" signified those participants who were evaluable for a specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 187 | 187
units on a scale
  Baseline | 22.58 (5.23) | 22.76 (4.61)
  CFB at Cycle 3 Day 1: number analyzed (Participants) | 156 | 154
  CFB at Cycle 3 Day 1 | -1.56 (5.49) | -0.69 (4.06)
  CFB at Cycle 4 Day 1: number analyzed (Participants) | 5 | 2
  CFB at Cycle 4 Day 1 | -6.80 (4.21) | -3.00 (2.83)
  CFB at Cycle 5 Day 1: number analyzed (Participants) | 142 | 145
  CFB at Cycle 5 Day 1 | -1.82 (5.06) | -0.72 (4.16)
  CFB at End of Induction Treatment: number analyzed (Participants) | 149 | 142
  CFB at End of Induction Treatment | -1.00 (5.14) | -0.61 (4.62)
  CFB at Follow-up Month 2: number analyzed (Participants) | 108 | 133
  CFB at Follow-up Month 2 | 0.62 (5.14) | 0.58 (4.45)
  CFB at Follow-up Month 4: number analyzed (Participants) | 95 | 121
  CFB at Follow-up Month 4 | 0.53 (4.58) | 0.88 (4.47)
  CFB at Follow-up Month 6: number analyzed (Participants) | 77 | 112
  CFB at Follow-up Month 6 | 0.29 (3.74) | 0.91 (3.82)
  CFB at Follow-up Month 8: number analyzed (Participants) | 75 | 104
  CFB at Follow-up Month 8 | -0.01 (3.53) | 0.87 (3.96)
  CFB at Follow-up Month 10: number analyzed (Participants) | 58 | 91
  CFB at Follow-up Month 10 | 0.06 (4.16) | 0.56 (3.81)
  CFB at Follow-up Month 12: number analyzed (Participants) | 53 | 90
  CFB at Follow-up Month 12 | 0.26 (4.02) | 0.74 (4.24)
  CFB at Follow-up Month 14: number analyzed (Participants) | 46 | 85
  CFB at Follow-up Month 14 | 0.03 (4.14) | 0.71 (3.94)
  CFB at Follow-up Month 16: number analyzed (Participants) | 42 | 82
  CFB at Follow-up Month 16 | -0.10 (3.49) | 1.31 (3.68)
  CFB at Follow-up Month 18: number analyzed (Participants) | 41 | 76
  CFB at Follow-up Month 18 | -0.22 (3.64) | 0.92 (3.99)
  CFB at Follow-up Month 20: number analyzed (Participants) | 34 | 73
  CFB at Follow-up Month 20 | -0.36 (3.70) | 0.74 (3.69)
  CFB at Follow-up Month 22: number analyzed (Participants) | 29 | 71
  CFB at Follow-up Month 22 | -0.25 (3.93) | 0.40 (4.47)
  CFB at Follow-up Month 24: number analyzed (Participants) | 30 | 68
  CFB at Follow-up Month 24 | -0.77 (4.16) | 0.52 (4.42)
  CFB at Final Follow-up: number analyzed (Participants) | 86 | 106
  CFB at Final Follow-up | 0.16 (4.17) | 0.22 (4.47)
  CFB at Extension Follow-up Month 6: number analyzed (Participants) | 21 | 60
  CFB at Extension Follow-up Month 6 | 0.36 (3.48) | 0.57 (4.71)
  CFB at Extension Follow-up Month 18: number analyzed (Participants) | 19 | 46
  CFB at Extension Follow-up Month 18 | 0.80 (2.54) | 1.19 (4.98)
  CFB at Extension Follow-up Month 24: number analyzed (Participants) | 18 | 39
  CFB at Extension Follow-up Month 24 | 1.53 (5.96) | 0.56 (5.26)

21. Secondary Outcome: CFB in FACT-Lym-Social/Family Well-being Sub-scale Score
Description: The FACT-Lym measures 5 sub-scales which includes 42 items; responses to each item range from 0, "Not at all" to 4, "Very much". Total score ranges from 0-168. Social/family Well-being sub-scale includes 7 items measured on 0-4 point scale. The total score for social/family well-being sub-scale is sum of each 7 items (range: 0-28). Higher scores indicate a better PRO/QoL. In timeframe, follow-up months represents months after end of induction (e.g. Follow-up Month 2 is 2 months after end of induction) and extension follow-up months represents months after end of 2 years normal follow-up (e.g. extension follow-up Month 6 is 6 months after end of normal 2 year follow-up).
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 186 | 191
units on a scale
  Baseline | 22.04 (5.65) | 22.14 (5.51)
  CFB at Cycle 3 Day 1: number analyzed (Participants) | 155 | 158
  CFB at Cycle 3 Day 1 | -0.21 (3.59) | -0.10 (3.87)
  CFB at Cycle 4 Day 1: number analyzed (Participants) | 5 | 3
  CFB at Cycle 4 Day 1 | -1.00 (3.67) | 3.11 (2.83)
  CFB at Cycle 5 Day 1: number analyzed (Participants) | 141 | 149
  CFB at Cycle 5 Day 1 | -0.34 (4.32) | -0.34 (4.33)
  CFB at End of Induction Treatment: number analyzed (Participants) | 147 | 145
  CFB at End of Induction Treatment | -0.65 (5.21) | -0.88 (3.60)
  CFB at Follow-up Month 2: number analyzed (Participants) | 106 | 137
  CFB at Follow-up Month 2 | -0.02 (4.83) | -0.57 (5.37)
  CFB at Follow-up Month 4: number analyzed (Participants) | 94 | 125
  CFB at Follow-up Month 4 | 0.27 (4.65) | -0.26 (5.02)
  CFB at Follow-up Month 6: number analyzed (Participants) | 76 | 114
  CFB at Follow-up Month 6 | 0.05 (4.46) | -0.08 (4.64)
  CFB at Follow-up Month 8 | -0.68 (3.67) | -0.37 (4.99)
  CFB at Follow-up Month 10: number analyzed (Participants) | 58 | 94
  CFB at Follow-up Month 10 | 0.56 (5.00) | 0.13 (5.14)
  CFB at Follow-up Month 12: number analyzed (Participants) | 53 | 93
  CFB at Follow-up Month 12 | 0.06 (5.89) | -0.47 (5.64)
  CFB at Follow-up Month 14: number analyzed (Participants) | 45 | 89
  CFB at Follow-up Month 14 | 0.56 (3.28) | -0.03 (4.16)
  CFB at Follow-up Month 16: number analyzed (Participants) | 42 | 85
  CFB at Follow-up Month 16 | 0.36 (6.79) | -0.15 (5.28)
  CFB at Follow-up Month 18: number analyzed (Participants) | 41 | 78
  CFB at Follow-up Month 18 | 0.44 (6.23) | 0.04 (5.35)
  CFB at Follow-up Month 20: number analyzed (Participants) | 34 | 76
  CFB at Follow-up Month 20 | -0.66 (4.28) | 0.00 (5.75)
  CFB at Follow-up Month 22: number analyzed (Participants) | 29 | 74
  CFB at Follow-up Month 22 | 0.29 (7.12) | -0.50 (5.02)
  CFB at Follow-up Month 24: number analyzed (Participants) | 30 | 71
  CFB at Follow-up Month 24 | -1.29 (3.91) | -0.41 (5.24)
  CFB at Final Follow-up: number analyzed (Participants) | 86 | 109
  CFB at Final Follow-up | -0.19 (4.91) | -0.52 (5.56)
  CFB at Extension Follow-up Month 6: number analyzed (Participants) | 21 | 63
  CFB at Extension Follow-up Month 6 | -0.35 (2.49) | -0.16 (4.92)
  CFB at Extension Follow-up Month 18: number analyzed (Participants) | 18 | 49
  CFB at Extension Follow-up Month 18 | -0.15 (2.92) | 0.71 (5.26)
  CFB at Extension Follow-up Month 24: number analyzed (Participants) | 18 | 40
  CFB at Extension Follow-up Month 24 | -0.41 (3.18) | 0.44 (5.02)

22. Secondary Outcome: CFB in FACT-Lym-Emotional Well-Being Sub-scale Score
Description: The FACT-Lym measures 5 sub-scales which includes 42 items; responses to each item range from 0, "Not at all" to 4, "Very much". Total score ranges from 0-168. Emotional Well-being sub-scale includes 6 items measured on 0-4 point scale. The total score for emotional well-being sub-scale is sum of each 6 items (range: 0-24). Higher scores indicate a better PRO/QoL. In timeframe, follow-up months represents months after end of induction (e.g. Follow-up Month 2 is 2 months after end of induction) and extension follow-up months represents months after end of 2 years normal follow-up (e.g. extension follow-up Month 6 is 6 months after end of normal 2 year follow-up).
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 189 | 193
units on a scale
  Baseline | 17.38 (4.45) | 17.81 (4.33)
  CFB at Cycle 3 Day 1: number analyzed (Participants) | 157 | 163
  CFB at Cycle 3 Day 1 | 0.61 (3.04) | 0.78 (3.14)
  CFB at Cycle 4 Day 1: number analyzed (Participants) | 5 | 3
  CFB at Cycle 4 Day 1 | -0.60 (3.85) | 3.40 (4.42)
  CFB at Cycle 5 Day 1: number analyzed (Participants) | 143 | 152
  CFB at Cycle 5 Day 1 | 0.37 (3.08) | 0.50 (3.52)
  CFB at End of Induction Treatment: number analyzed (Participants) | 149 | 145
  CFB at End of Induction Treatment | 0.53 (3.57) | 0.59 (4.03)
  CFB at Follow-up Month 2: number analyzed (Participants) | 107 | 138
  CFB at Follow-up Month 2 | 0.66 (3.89) | 0.67 (3.83)
  CFB at Follow-up Month 4: number analyzed (Participants) | 96 | 124
  CFB at Follow-up Month 4 | 1.34 (3.54) | 0.95 (3.51)
  CFB at Follow-up Month 6: number analyzed (Participants) | 78 | 116
  CFB at Follow-up Month 6 | 0.89 (3.57) | 0.96 (3.44)
  CFB at Follow-up Month 8: number analyzed (Participants) | 76 | 108
  CFB at Follow-up Month 8 | 0.26 (3.35) | 0.97 (3.34)
  CFB at Follow-up Month 10: number analyzed (Participants) | 58 | 94
  CFB at Follow-up Month 10 | 0.69 (3.31) | 1.32 (3.23)
  CFB at Follow-up Month 12: number analyzed (Participants) | 54 | 93
  CFB at Follow-up Month 12 | -0.07 (3.88) | 0.95 (3.29)
  CFB at Follow-up Month 14: number analyzed (Participants) | 47 | 89
  CFB at Follow-up Month 14 | 0.46 (3.22) | 1.07 (3.82)
  CFB at Follow-up Month 16: number analyzed (Participants) | 43 | 86
  CFB at Follow-up Month 16 | 0.13 (3.87) | 1.04 (3.69)
  CFB at Follow-up Month 18: number analyzed (Participants) | 41 | 79
  CFB at Follow-up Month 18 | 0.42 (3.36) | 1.00 (3.38)
  CFB at Follow-up Month 20: number analyzed (Participants) | 35 | 76
  CFB at Follow-up Month 20 | -0.43 (2.90) | 0.94 (4.28)
  CFB at Follow-up Month 22: number analyzed (Participants) | 30 | 74
  CFB at Follow-up Month 22 | 0.18 (2.81) | 0.97 (3.79)
  CFB at Follow-up Month 24: number analyzed (Participants) | 31 | 71
  CFB at Follow-up Month 24 | 0.06 (3.20) | 1.12 (3.78)
  CFB at Final Follow-up: number analyzed (Participants) | 84 | 111
  CFB at Final Follow-up | 0.38 (3.77) | 0.34 (4.37)
  CFB at Extension Follow-up Month 6: number analyzed (Participants) | 23 | 63
  CFB at Extension Follow-up Month 6 | -0.44 (3.26) | 0.39 (3.99)
  CFB at Extension Follow-up Month 18: number analyzed (Participants) | 20 | 50
  CFB at Extension Follow-up Month 18 | -0.08 (3.80) | 0.75 (3.85)
  CFB at Extension Follow-up Month 24: number analyzed (Participants) | 19 | 42
  CFB at Extension Follow-up Month 24 | 1.04 (4.16) | 0.97 (4.36)

23. Secondary Outcome: CFB in FACT-Lym-Functional Well-Being Sub-scale Score
Description: The FACT-Lym measures 5 sub-scales which includes 42 items; responses to each item range from 0, "Not at all" to 4, "Very much". Total score ranges from 0-168. Functional Well-being sub-scale includes 7 items measured on 0-4 point scale. The total score for functional well-being sub-scale is sum of each 7 items (range: 0-28). Higher scores indicate a better PRO/QoL. In timeframe, follow-up months represents months after end of induction (e.g. Follow-up Month 2 is 2 months after end of induction) and extension follow-up months represents months after end of 2 years normal follow-up (e.g. extension follow-up Month 6 is 6 months after end of normal 2 year follow-up).
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 189 | 196
units on a scale
  Baseline | 17.98 (6.31) | 17.90 (6.08)
  CFB at Cycle 3 Day 1: number analyzed (Participants) | 157 | 165
  CFB at Cycle 3 Day 1 | -0.54 (4.65) | 0.38 (4.66)
  CFB at Cycle 4 Day 1: number analyzed (Participants) | 5 | 3
  CFB at Cycle 4 Day 1 | -0.80 (2.28) | 1.78 (4.91)
  CFB at Cycle 5 Day 1: number analyzed (Participants) | 143 | 154
  CFB at Cycle 5 Day 1 | -0.71 (5.04) | 0.67 (5.35)
  CFB at End of Induction Treatment: number analyzed (Participants) | 150 | 147
  CFB at End of Induction Treatment | -0.50 (5.50) | 0.00 (5.25)
  CFB at Follow-up Month 2: number analyzed (Participants) | 107 | 139
  CFB at Follow-up Month 2 | 0.31 (5.27) | 0.65 (5.38)
  CFB at Follow-up Month 4: number analyzed (Participants) | 96 | 126
  CFB at Follow-up Month 4 | 0.24 (5.11) | 1.31 (5.86)
  CFB at Follow-up Month 6: number analyzed (Participants) | 77 | 117
  CFB at Follow-up Month 6 | 0.95 (4.58) | 1.26 (5.08)
  CFB at Follow-up Month 8: number analyzed (Participants) | 76 | 109
  CFB at Follow-up Month 8 | -0.27 (4.38) | 0.92 (5.45)
  CFB at Follow-up Month 10: number analyzed (Participants) | 59 | 96
  CFB at Follow-up Month 10 | 1.09 (4.25) | 1.00 (5.52)
  CFB at Follow-up Month 12: number analyzed (Participants) | 54 | 95
  CFB at Follow-up Month 12 | 0.18 (5.59) | 1.78 (6.04)
  CFB at Follow-up Month 14: number analyzed (Participants) | 47 | 90
  CFB at Follow-up Month 14 | 1.16 (4.27) | 1.22 (4.84)
  CFB at Follow-up Month 16: number analyzed (Participants) | 43 | 87
  CFB at Follow-up Month 16 | 0.91 (3.97) | 1.69 (5.95)
  CFB at Follow-up Month 18: number analyzed (Participants) | 41 | 79
  CFB at Follow-up Month 18 | 0.21 (4.12) | 1.84 (5.77)
  CFB at Follow-up Month 20: number analyzed (Participants) | 35 | 77
  CFB at Follow-up Month 20 | -0.27 (4.90) | 1.43 (6.14)
  CFB at Follow-up Month 22: number analyzed (Participants) | 30 | 75
  CFB at Follow-up Month 22 | -0.32 (5.70) | 0.82 (5.00)
  CFB at Follow-up Month 24: number analyzed (Participants) | 31 | 71
  CFB at Follow-up Month 24 | -0.96 (4.36) | 0.98 (5.87)
  CFB at Final Follow-up: number analyzed (Participants) | 84 | 114
  CFB at Final Follow-up | -0.08 (4.94) | 0.50 (6.19)
  CFB at Extension Follow-up Month 6: number analyzed (Participants) | 23 | 63
  CFB at Extension Follow-up Month 6 | 1.01 (3.51) | 0.85 (6.65)
  CFB at Extension Follow-up Month 18: number analyzed (Participants) | 19 | 50
  CFB at Extension Follow-up Month 18 | 0.96 (4.51) | 1.90 (6.50)
  CFB at Extension Follow-up Month 24: number analyzed (Participants) | 19 | 42
  CFB at Extension Follow-up Month 24 | 2.22 (3.34) | 2.62 (6.95)

24. Secondary Outcome: CFB in FACT-Lym-Lymphoma Sub-scale Score
Description: The FACT-Lym measures 5 sub-scales which includes 42 items; responses to each item range from 0, "Not at all" to 4, "Very much". Total score ranges from 0-168. Lymphoma scale includes 15 items measured on 0-4 point scale. The total score for lymphoma sub-scale is sum of each 15 items (range: 0-60). Higher scores indicate a better PRO/QoL. In timeframe, follow-up months represents months after end of induction (e.g. Follow-up Month 2 is 2 months after end of induction) and extension follow-up months represents months after end of 2 years normal follow-up (e.g. extension follow-up Month 6 is 6 months after end of normal 2 year follow-up).
Time Frame: as for outcome 20
Population: ITT population. Here, number of participants analyzed signified those participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 189 | 194
units on a scale
  Baseline | 44.79 (9.66) | 45.61 (9.17)
  CFB at Cycle 3 Day 1: number analyzed (Participants) | 154 | 162
  CFB at Cycle 3 Day 1 | 0.98 (6.97) | 1.24 (5.71)
  CFB at Cycle 4 Day 1: number analyzed (Participants) | 5 | 2
  CFB at Cycle 4 Day 1 | -2.80 (5.76) | 9.50 (3.54)
  CFB at Cycle 5 Day 1: number analyzed (Participants) | 142 | 151
  CFB at Cycle 5 Day 1 | 0.75 (6.79) | 1.41 (6.21)
  CFB at End of Induction Treatment: number analyzed (Participants) | 148 | 148
  CFB at End of Induction Treatment | 1.64 (7.10) | 0.74 (7.89)
  CFB at Follow-up Month 2: number analyzed (Participants) | 107 | 135
  CFB at Follow-up Month 2 | 3.44 (6.78) | 2.45 (6.22)
  CFB at Follow-up Month 4: number analyzed (Participants) | 96 | 123
  CFB at Follow-up Month 4 | 2.77 (6.71) | 2.39 (6.54)
  CFB at Follow-up Month 6: number analyzed (Participants) | 79 | 117
  CFB at Follow-up Month 6 | 2.33 (6.44) | 3.00 (7.05)
  CFB at Follow-up Month 8: number analyzed (Participants) | 75 | 107
  CFB at Follow-up Month 8 | 1.79 (6.01) | 2.52 (6.69)
  CFB at Follow-up Month 10: number analyzed (Participants) | 59 | 94
  CFB at Follow-up Month 10 | 1.90 (6.78) | 2.28 (6.82)
  CFB at Follow-up Month 12: number analyzed (Participants) | 53 | 94
  CFB at Follow-up Month 12 | 2.12 (6.47) | 2.89 (6.42)
  CFB at Follow-up Month 14: number analyzed (Participants) | 47 | 91
  CFB at Follow-up Month 14 | 0.48 (6.64) | 2.58 (6.37)
  CFB at Follow-up Month 16: number analyzed (Participants) | 42 | 86
  CFB at Follow-up Month 16 | 0.44 (7.79) | 3.27 (6.14)
  CFB at Follow-up Month 18: number analyzed (Participants) | 42 | 78
  CFB at Follow-up Month 18 | 1.18 (6.09) | 2.91 (6.79)
  CFB at Follow-up Month 20: number analyzed (Participants) | 34 | 75
  CFB at Follow-up Month 20 | 0.57 (7.43) | 2.83 (6.41)
  CFB at Follow-up Month 22: number analyzed (Participants) | 30 | 72
  CFB at Follow-up Month 22 | 1.89 (8.62) | 2.55 (6.58)
  CFB at Follow-up Month 24: number analyzed (Participants) | 31 | 70
  CFB at Follow-up Month 24 | 0.66 (7.59) | 2.73 (6.48)
  CFB at Final Follow-up: number analyzed (Participants) | 85 | 112
  CFB at Final Follow-up | 1.62 (7.17) | 1.33 (7.38)
  CFB at Extension Follow-up Month 6: number analyzed (Participants) | 23 | 61
  CFB at Extension Follow-up Month 6 | 0.92 (5.06) | 2.98 (7.22)
  CFB at Extension Follow-up Month 18: number analyzed (Participants) | 20 | 50
  CFB at Extension Follow-up Month 18 | 1.80 (8.30) | 2.35 (5.72)
  CFB at Extension Follow-up Month 24: number analyzed (Participants) | 19 | 42
  CFB at Extension Follow-up Month 24 | 4.89 (6.67) | 2.23 (6.85)

25. Secondary Outcome: CFB in Euro Quality of Life 5 Dimension (EuroQoL-5D/EQ-5D) - Health State Profile Utility Score During Induction Phase
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQoL Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state. In timeframe, follow-up months represents months after end of induction (e.g. Follow-up Month 2 is 2 months after end of induction). For 'Obinutuzumab + Bendamustine' arm, participants who had their follow-up Month 2 and 4 visits before start of maintenance treatment were reported in induction phase results under "CFB at Follow-up Month 2" and "CFB at Follow-up Month 4" categories.
Time Frame: Baseline, Day 1 of Cycles 3, 4, 5, End of induction treatment (up to Month 6); Follow-up Months 2, 4 and 14
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 186 | 193
units on a scale
  Baseline | 0.77 (0.22) | 0.79 (0.20)
  CFB at Cycle 3 Day 1: number analyzed (Participants) | 157 | 161
  CFB at Cycle 3 Day 1 | 0.03 (0.21) | 0.00 (0.19)
  CFB at Cycle 4 Day 1: number analyzed (Participants) | 5 | 3
  CFB at Cycle 4 Day 1 | -0.10 (0.23) | -0.07 (0.41)
  CFB at Cycle 5 Day 1: number analyzed (Participants) | 142 | 153
  CFB at Cycle 5 Day 1 | 0.01 (0.21) | 0.02 (0.20)
  CFB at End of Induction Treatment: number analyzed (Participants) | 136 | 140
  CFB at End of Induction Treatment | 0.01 (0.22) | 0.01 (0.20)
  CFB at Follow-up Month 2: number analyzed (Participants) | 39 | 135
  CFB at Follow-up Month 2 | 0.06 (0.24) | 0.04 (0.18)
  CFB at Follow-up Month 4: number analyzed (Participants) | 0 | 2
  CFB at Follow-up Month 4 |  | -0.12 (0.00)
  CFB at Follow-up Month 14: number analyzed (Participants) | 1 | 0
  CFB at Follow-up Month 14 | 0.12 (NA) — Standard deviation is non-evaluable due to low number of participants. |

26. Secondary Outcome: CFB in EuroQol 5D (EQ-5D) - Health State Profile Utility Score During Maintenance Phase
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQoL Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state. Data for this outcome was planned to be reported only for 'Obinutuzumab + Bendamustine' arm. In timeframe, follow-up months represents months after end of induction (e.g. Follow-up Month 2 is 2 months after end of induction). Follow-up months were during maintenance phase.
Time Frame: Baseline, Follow-up Months 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, Final follow-up (up to 2 years after end of induction) (End of induction = up to Month 6)
Population: ITT population (Obinutuzumab + Bendamustine arm only). Here, number of participants analyzed signified those participants who were evaluable for this outcome and "n" signified those participants who were evaluable for a specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 2 | 158
units on a scale
  CFB at Follow-up Month 2: number analyzed (Participants) | 0 | 2
  CFB at Follow-up Month 2 |  | -0.15 (0.22)
  CFB at Follow-up Month 4: number analyzed (Participants) | 1 | 119
  CFB at Follow-up Month 4 | 0.15 (NA) — Standard deviation was not evaluable due to low number of participants. | 0.03 (0.22)
  CFB at Follow-up Month 6: number analyzed (Participants) | 1 | 109
  CFB at Follow-up Month 6 | 0.15 (NA) — Standard deviation was not evaluable due to low number of participants. | 0.04 (0.19)
  CFB at Follow-up Month 8: number analyzed (Participants) | 1 | 101
  CFB at Follow-up Month 8 | 0.15 (NA) — Standard deviation is non-evaluable due to low number of participants. | 0.04 (0.21)
  CFB at Follow-up Month 10: number analyzed (Participants) | 1 | 91
  CFB at Follow-up Month 10 | 0.15 (NA) — Standard deviation was not evaluable due to low number of participants. | 0.03 (0.20)
  CFB at Follow-up Month 12: number analyzed (Participants) | 0 | 87
  CFB at Follow-up Month 12 |  | 0.06 (0.18)
  CFB at Follow-up Month 14: number analyzed (Participants) | 0 | 80
  CFB at Follow-up Month 14 |  | 0.06 (0.19)
  CFB at Follow-up Month 16: number analyzed (Participants) | 0 | 78
  CFB at Follow-up Month 16 |  | 0.05 (0.19)
  CFB at Follow-up Month 18: number analyzed (Participants) | 0 | 73
  CFB at Follow-up Month 18 |  | 0.05 (0.18)
  CFB at Follow-up Month 20: number analyzed (Participants) | 0 | 69
  CFB at Follow-up Month 20 |  | 0.05 (0.20)
  CFB at Follow-up Month 22: number analyzed (Participants) | 0 | 69
  CFB at Follow-up Month 22 |  | 0.05 (0.24)
  CFB at Follow-up Month 24: number analyzed (Participants) | 0 | 64
  CFB at Follow-up Month 24 |  | 0.03 (0.22)
  CFB at Final Follow-up: number analyzed (Participants) | 0 | 39
  CFB at Final Follow-up |  | 0.03 (0.25)

27. Secondary Outcome: CFB in EQ-5D Visual Analogue Scale (VAS) Score During Induction Phase
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 millimeter (mm) (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state. In timeframe, follow-up months represents months after end of induction (e.g. Follow-up Month 2 is 2 months after end of induction). For 'Obinutuzumab + Bendamustine' arm, participants who had their follow-up Month 2 and 4 visits before start of maintenance treatment were reported in induction phase results under "CFB at Follow-up Month 2" and "CFB at Follow-up Month 4" categories.
Time Frame: Baseline, Day 1 of Cycles 3, 4, 5, End of induction treatment (up to Month 6); Follow-up Months 2, 4 and 14
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 183 | 188
units on a scale
  Baseline | 69.48 (20.71) | 68.03 (21.69)
  CFB at Cycle 3 Day 1: number analyzed (Participants) | 152 | 153
  CFB at Cycle 3 Day 1 | 0.91 (19.38) | 3.32 (15.99)
  CFB at Cycle 4 Day 1: number analyzed (Participants) | 5 | 3
  CFB at Cycle 4 Day 1 | -14.00 (33.29) | -4.33 (42.15)
  CFB at Cycle 5 Day 1: number analyzed (Participants) | 136 | 141
  CFB at Cycle 5 Day 1 | 0.35 (20.79) | 5.17 (17.35)
  CFB at End of Induction Treatment: number analyzed (Participants) | 132 | 135
  CFB at End of Induction Treatment | 5.71 (61.88) | 5.82 (22.20)
  CFB at Follow-up Month 2: number analyzed (Participants) | 36 | 128
  CFB at Follow-up Month 2 | 5.19 (19.12) | 6.85 (18.95)
  CFB at Follow-up Month 4: number analyzed (Participants) | 0 | 2
  CFB at Follow-up Month 4 |  | 0.00 (14.14)
  CFB at Follow-up Month 14: number analyzed (Participants) | 1 | 0
  CFB at Follow-up Month 14 | 10.00 (NA) — Standard deviation is non-evaluable due to low number of participants. |

28. Secondary Outcome: CFB in EQ-5D VAS Score During Maintenance Phase
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 mm (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state. Data for this outcome was planned to be reported only for 'Obinutuzumab + Bendamustine' arm. In timeframe, follow-up months represents months after end of induction (e.g. Follow-up Month 2 is 2 months after end of induction). Follow-up months were during maintenance phase.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 2 | 158
units on a scale
  CFB at Follow-up Month 2: number analyzed (Participants) | 0 | 1
  CFB at Follow-up Month 2 |  | -40.00 (NA) — SD data not applicable as only one participant was evaluable for this time point.
  CFB at Follow-up Month 4: number analyzed (Participants) | 1 | 111
  CFB at Follow-up Month 4 | 5.00 (NA) — SD data not applicable as only one participant was evaluable for this time point. | 5.59 (19.61)
  CFB at Follow-up Month 6: number analyzed (Participants) | 1 | 106
  CFB at Follow-up Month 6 | 5.00 (NA) — SD data not applicable as only one participant was evaluable for this time point. | 6.04 (19.00)
  CFB at Follow-up Month 8: number analyzed (Participants) | 1 | 95
  CFB at Follow-up Month 8 | 5.00 (NA) — SD data not applicable as only one participant was evaluable for this time point. | 4.79 (17.18)
  CFB at Follow-up Month 10: number analyzed (Participants) | 1 | 86
  CFB at Follow-up Month 10 | -15.00 (NA) — SD data not applicable as only one participant was evaluable for this time point. | 4.62 (16.28)
  CFB at Follow-up Month 12: number analyzed (Participants) | 0 | 82
  CFB at Follow-up Month 12 |  | 5.73 (16.04)
  CFB at Follow-up Month 14: number analyzed (Participants) | 0 | 77
  CFB at Follow-up Month 14 |  | 5.45 (17.36)
  CFB at Follow-up Month 16: number analyzed (Participants) | 0 | 76
  CFB at Follow-up Month 16 |  | 6.66 (17.44)
  CFB at Follow-up Month 18: number analyzed (Participants) | 0 | 69
  CFB at Follow-up Month 18 |  | 6.13 (19.44)
  CFB at Follow-up Month 20: number analyzed (Participants) | 0 | 66
  CFB at Follow-up Month 20 |  | 7.56 (15.43)
  CFB at Follow-up Month 22: number analyzed (Participants) | 0 | 64
  CFB at Follow-up Month 22 |  | 6.97 (15.55)
  CFB at Follow-up Month 24: number analyzed (Participants) | 0 | 61
  CFB at Follow-up Month 24 |  | 8.28 (16.23)
  CFB at Final Follow-up: number analyzed (Participants) | 0 | 38
  CFB at Final Follow-up |  | 4.47 (14.91)

29. Secondary Outcome: CFB in Functional Assessment of Cancer Therapy - Generic (FACT-G) Score
Description: The FACT-G is the sum of 4 sub-scales (physical, social, emotional and functional well-being) of FACT-Lym which includes total 27 items; responses to each item range from 0, "Not at all" to 4, "Very much". Total score ranges from 0-108. Higher scores indicate a better PRO/QoL. In timeframe, follow-up months represents months after end of induction (e.g. Follow-up Month 2 is 2 months after end of induction) and extension follow-up months represents months after end of 2 years normal follow-up (e.g. extension follow-up Month 6 is 6 months after end of normal 2 year follow-up).
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 185 | 186
Units on a scale
  Baseline | 79.86 (16.25) | 80.78 (16.27)
  CFB at Cycle 3 Day 1: number analyzed (Participants) | 154 | 154
  CFB at Cycle 3 Day 1 | -1.87 (12.28) | 0.11 (10.30)
  CFB at Cycle 4 Day 1: number analyzed (Participants) | 5 | 2
  CFB at Cycle 4 Day 1 | -9.37 (9.89) | 0.52 (4.98)
  CFB at Cycle 5 Day 1: number analyzed (Participants) | 140 | 145
  CFB at Cycle 5 Day 1 | -2.44 (12.01) | 0.06 (11.13)
  CFB at End of Induction Treatment: number analyzed (Participants) | 146 | 140
  CFB at End of Induction Treatment | -1.84 (13.83) | -0.92 (11.77)
  CFB at Follow-up Month 2: number analyzed (Participants) | 107 | 133
  CFB at Follow-up Month 2 | 1.53 (13.42) | 1.22 (12.01)
  CFB at Follow-up Month 4: number analyzed (Participants) | 95 | 120
  CFB at Follow-up Month 4 | 2.55 (11.47) | 3.06 (13.00)
  CFB at Follow-up Month 6: number analyzed (Participants) | 75 | 111
  CFB at Follow-up Month 6 | 2.54 (10.68) | 3.24 (11.40)
  CFB at Follow-up Month 8: number analyzed (Participants) | 74 | 104
  CFB at Follow-up Month 8 | -0.53 (10.15) | 2.49 (11.45)
  CFB at Follow-up Month 10: number analyzed (Participants) | 57 | 88
  CFB at Follow-up Month 10 | 2.29 (11.39) | 3.46 (11.83)
  CFB at Follow-up Month 12: number analyzed (Participants) | 53 | 90
  CFB at Follow-up Month 12 | 0.68 (13.16) | 2.82 (14.29)
  CFB at Follow-up Month 14: number analyzed (Participants) | 45 | 84
  CFB at Follow-up Month 14 | 2.48 (9.42) | 2.94 (11.97)
  CFB at Follow-up Month 16: number analyzed (Participants) | 42 | 82
  CFB at Follow-up Month 16 | 1.54 (10.61) | 4.09 (12.87)
  CFB at Follow-up Month 18: number analyzed (Participants) | 39 | 76
  CFB at Follow-up Month 18 | 1.16 (11.57) | 4.06 (13.36)
  CFB at Follow-up Month 20: number analyzed (Participants) | 33 | 73
  CFB at Follow-up Month 20 | -1.21 (12.25) | 3.05 (14.29)
  CFB at Follow-up Month 22: number analyzed (Participants) | 28 | 71
  CFB at Follow-up Month 22 | 0.64 (14.27) | 1.80 (12.43)
  CFB at Follow-up Month 24: number analyzed (Participants) | 29 | 67
  CFB at Follow-up Month 24 | -2.39 (9.32) | 2.28 (13.83)
  CFB at Final Follow-up: number analyzed (Participants) | 84 | 106
  CFB at Final Follow-up | 0.50 (11.25) | 0.78 (14.94)
  CFB at Extension Follow Up Month 6: number analyzed (Participants) | 21 | 60
  CFB at Extension Follow Up Month 6 | 0.48 (8.71) | 1.74 (14.23)
  CFB at Extension Follow Up Month 18: number analyzed (Participants) | 18 | 46
  CFB at Extension Follow Up Month 18 | 2.29 (8.40) | 4.56 (15.02)
  CFB at Extension Follow Up Month 24: number analyzed (Participants) | 18 | 38
  CFB at Extension Follow Up Month 24 | 4.48 (11.10) | 4.47 (15.22)

30. Secondary Outcome: CFB in FACT-Lym Trial Outcome Index (TOI)
Description: TOI is the sum of 3 sub-scales (physical well-being, functional well-being, and Lymphoma sub-scale) of FACT-Lym which includes total 29 items; responses to each item range from 0, "Not at all" to 4, "Very much". Total score ranges from 0-116. Higher scores indicate a better PRO/QoL. In timeframe, follow-up months represents months after end of induction (e.g. Follow-up Month 2 is 2 months after end of induction) and extension follow-up months represents months after end of 2 years normal follow-up (e.g. extension follow-up Month 6 is 6 months after end of normal 2 year follow-up).
Time Frame: as for outcome 20
Population: ITT population. Here, number of participants analyzed signified those participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 190 | 196
Units on a scale
  Baseline | 84.66 (19.36) | 84.76 (18.97)
  CFB at Cycle 3 Day 1: number analyzed (Participants) | 159 | 165
  CFB at Cycle 3 Day 1 | -1.94 (17.96) | 1.81 (13.88)
  CFB at Cycle 4 Day 1: number analyzed (Participants) | 5 | 3
  CFB at Cycle 4 Day 1 | -10.40 (10.38) | 26.44 (19.51)
  CFB at Cycle 5 Day 1: number analyzed (Participants) | 144 | 154
  CFB at Cycle 5 Day 1 | -1.38 (15.38) | 2.37 (14.15)
  CFB at End of Induction Treatment: number analyzed (Participants) | 151 | 149
  CFB at End of Induction Treatment | -0.52 (17.23) | 0.40 (16.45)
  CFB at Follow-up Month 2: number analyzed (Participants) | 108 | 139
  CFB at Follow-up Month 2 | 3.75 (15.36) | 4.60 (14.85)
  CFB at Follow-up Month 4: number analyzed (Participants) | 96 | 127
  CFB at Follow-up Month 4 | 3.81 (13.39) | 5.18 (17.06)
  CFB at Follow-up Month 6: number analyzed (Participants) | 79 | 117
  CFB at Follow-up Month 6 | 3.26 (12.19) | 6.07 (13.72)
  CFB at Follow-up Month 8: number analyzed (Participants) | 76 | 109
  CFB at Follow-up Month 8 | 1.36 (12.39) | 5.36 (14.21)
  CFB at Follow-up Month 10: number analyzed (Participants) | 59 | 96
  CFB at Follow-up Month 10 | 3.52 (13.16) | 4.94 (15.96)
  CFB at Follow-up Month 12: number analyzed (Participants) | 54 | 95
  CFB at Follow-up Month 12 | 2.05 (15.14) | 6.13 (15.72)
  CFB at Follow-up Month 14: number analyzed (Participants) | 47 | 91
  CFB at Follow-up Month 14 | 2.25 (11.92) | 5.13 (14.30)
  CFB at Follow-up Month 16: number analyzed (Participants) | 43 | 87
  CFB at Follow-up Month 16 | 0.75 (14.15) | 6.78 (15.11)
  CFB at Follow-up Month 18: number analyzed (Participants) | 42 | 79
  CFB at Follow-up Month 18 | 1.36 (11.30) | 7.26 (14.62)
  CFB at Follow-up Month 20: number analyzed (Participants) | 35 | 77
  CFB at Follow-up Month 20 | -0.64 (15.21) | 6.36 (14.99)
  CFB at Follow-up Month 22: number analyzed (Participants) | 30 | 75
  CFB at Follow-up Month 22 | 2.26 (14.54) | 5.30 (17.88)
  CFB at Follow-up Month 24: number analyzed (Participants) | 31 | 72
  CFB at Follow-up Month 24 | -0.14 (13.44) | 5.30 (17.88)
  CFB at Final Follow-up: number analyzed (Participants) | 86 | 114
  CFB at Final Follow-up | 0.84 (14.80) | 3.84 (16.22)
  CFB at Extension Follow Up Month 6: number analyzed (Participants) | 23 | 63
  CFB at Extension Follow Up Month 6 | 2.30 (10.77) | 5.53 (18.44)
  CFB at Extension Follow Up Month 18: number analyzed (Participants) | 20 | 50
  CFB at Extension Follow Up Month 18 | 4.02 (14.01) | 7.31 (15.69)
  CFB at Extension Follow Up Month 24: number analyzed (Participants) | 19 | 42
  CFB at Extension Follow Up Month 24 | 10.04 (13.35) | 7.07 (17.59)

31. Secondary Outcome: CFB in FACT-Lym Total Score
Description: FACT-Lym total score is the sum of physical well-being score (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and Lymphoma sub-scale (15 items); responses to each item range from 0, "Not at all" to 4, "Very much". Total score ranges from 0-168. Higher scores indicate a better PRO/QoL. In timeframe, follow-up months represents months after end of induction (e.g. Follow-up Month 2 is 2 months after end of induction) and extension follow-up months represents months after end of 2 years normal follow-up (e.g. extension follow-up Month 6 is 6 months after end of normal 2 year follow-up).
Time Frame: as for outcome 20
Population: ITT population. Here, number of participants analyzed signified those participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 186 | 187
Units on a scale
  Baseline | 124.56 (24.17) | 126.22 (23.98)
  CFB at Cycle 3 Day 1: number analyzed (Participants) | 153 | 154
  CFB at Cycle 3 Day 1 | -0.74 (17.91) | 1.33 (13.89)
  CFB at Cycle 4 Day 1: number analyzed (Participants) | 5 | 2
  CFB at Cycle 4 Day 1 | -12.16 (14.80) | 22.53 (16.23)
  CFB at Cycle 5 Day 1: number analyzed (Participants) | 140 | 144
  CFB at Cycle 5 Day 1 | -1.68 (16.61) | 1.71 (15.23)
  CFB at End of Induction Treatment: number analyzed (Participants) | 147 | 140
  CFB at End of Induction Treatment | 0.02 (18.55) | 0.35 (18.29)
  CFB at Follow-up Month 2: number analyzed (Participants) | 106 | 131
  CFB at Follow-up Month 2 | 5.10 (17.73) | 3.54 (15.45)
  CFB at Follow-up Month 4: number analyzed (Participants) | 95 | 119
  CFB at Follow-up Month 4 | 5.40 (16.29) | 5.50 (17.76)
  CFB at Follow-up Month 6: number analyzed (Participants) | 76 | 113
  CFB at Follow-up Month 6 | 5.03 (15.01) | 6.57 (15.96)
  CFB at Follow-up Month 8: number analyzed (Participants) | 74 | 104
  CFB at Follow-up Month 8 | 1.48 (14.27) | 5.18 (15.61)
  CFB at Follow-up Month 10: number analyzed (Participants) | 58 | 91
  CFB at Follow-up Month 10 | 4.58 (16.39) | 5.70 (16.89)
  CFB at Follow-up Month 12: number analyzed (Participants) | 52 | 91
  CFB at Follow-up Month 12 | 2.97 (17.84) | 5.88 (18.93)
  CFB at Follow-up Month 14: number analyzed (Participants) | 45 | 87
  CFB at Follow-up Month 14 | 3.18 (13.85) | 5.92 (17.06)
  CFB at Follow-up Month 16: number analyzed (Participants) | 41 | 83
  CFB at Follow-up Month 16 | 2.25 (14.98) | 7.59 (16.97)
  CFB at Follow-up Month 18: number analyzed (Participants) | 40 | 76
  CFB at Follow-up Month 18 | 2.16 (15.38) | 6.99 (18.27)
  CFB at Follow-up Month 20: number analyzed (Participants) | 33 | 73
  CFB at Follow-up Month 20 | -0.89 (16.34) | 5.66 (18.90)
  CFB at Follow-up Month 22: number analyzed (Participants) | 29 | 71
  CFB at Follow-up Month 22 | 2.15 (19.03) | 4.59 (17.98)
  CFB at Follow-up Month 24: number analyzed (Participants) | 30 | 67
  CFB at Follow-up Month 24 | -2.13 (15.74) | 5.28 (18.75)
  CFB at Final follow-up: number analyzed (Participants) | 84 | 105
  CFB at Final follow-up | 2.15 (16.60) | 2.55 (20.11)
  CFB at Extension Follow Up Month 6: number analyzed (Participants) | 21 | 60
  CFB at Extension Follow Up Month 6 | 1.22 (11.67) | 5.14 (20.30)
  CFB at Extension Follow Up Month 18: number analyzed (Participants) | 18 | 48
  CFB at Extension Follow Up Month 18 | 4.92 (14.73) | 6.88 (19.24)
  CFB at Extension Follow Up Month 24: number analyzed (Participants) | 18 | 41
  CFB at Extension Follow Up Month 24 | 9.69 (15.88) | 6.13 (20.32)

32. Secondary Outcome: Time to Deterioration of FACT-Lym TOI
Description: The median time, in month, from date of randomization until a clinically meaningful decline from baseline in TOI or death, whichever occurred first. TOI: sum of physical well-being score,functional well-being score, and Lymphoma sub-scale of FACT-Lym; total 29 items, responses to each item range from 0, "Not at all" to 4, "Very much". Total score ranges from 0-116. Higher scores indicate a better PRO/QoL. A clinically meaningful decline in TOI score was defined as at least a 6 point decline from baseline. Time to deterioration was estimated using Kaplan-Meier method and 95% CI for median was computed using the method of Brookmeyer and Crowley. In timeframe, follow-up months represents months after end of induction (EOI) (e.g. Follow-up Month 2 is 2 months after end of induction) and extension follow-up months represents months after end of 2 years normal follow-up (e.g. extension follow-up Month 6 is 6 months after end of normal 2 year follow-up).
Time Frame: Baseline up to approximately 8.5 years
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
Months | 5.6 [3.9 to 7.0] | 8.0 [5.9 to 14.7]

33. Secondary Outcome: Percentage of Participants With Definitive Improvement (DI) From Baseline in FACT-Lym Instrument Scores
Description: FACT-Lym: 42-items in 5 subscales. Responses to each item range from 0 (Not at all) to 4 (Very much). FACT-Lym Lymphoma subscale includes 15 items (total score range = 0-60). FACT-Lym TOI is sum of 3 subscales (physical well-being, functional well-being, lymphoma subscale) and includes 29 items (total score range = 0-116). FACT-Lym total score is sum of 42 items (total score ranges from 0-168). For all above, higher scores indicate a better PRO/QoL. DI from baseline: at least 3 point increase from baseline in FACT-Lym Lymphoma subscale; at least 6 point increase from baseline in FACT Lym TOI; at least 7 point increase from baseline in FACT Lym total scores. In timeframe, follow-up months represents months after EOI (e.g. Follow-up Month 2 is 2 months after EOI; EOI = up to Month 6).
Time Frame: Baseline, Cycle 5 Day 1 (C5D1) (Cycle length = 28 days), Follow-up Months 6 (FUM6), 12 (FUM12), 18 (FUM18), 24 (FUM24), Extension Follow Up Month 6 (Extension FUM6)
Population: ITT population. Here, number of participants analyzed signified those participants who were evaluable for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 209 | 204
Percentage of participants
  C5D1 (>=3 pt increase): number analyzed (Participants) | 155 | 156
  C5D1 (>=3 pt increase) | 30.3 | 41.7
  FUM6 (>=3 pt increase): number analyzed (Participants) | 87 | 119
  FUM6 (>=3 pt increase) | 37.9 | 47.1
  FUM12 (>=3 pt increase): number analyzed (Participants) | 60 | 99
  FUM12 (>=3 pt increase) | 36.7 | 46.5
  FUM18 (>=3 pt increase): number analyzed (Participants) | 45 | 83
  FUM18 (>=3 pt increase) | 35.6 | 53.0
  FUM24 (>=3 pt increase): number analyzed (Participants) | 34 | 74
  FUM24 (>=3 pt increase) | 35.3 | 50
  Ext FUM6 (>=3 pt increase): number analyzed (Participants) | 25 | 64
  Ext FUM6 (>=3 pt increase) | 36.0 | 57.8
  C5D1 (>=6 pt increase): number analyzed (Participants) | 156 | 157
  C5D1 (>=6 pt increase) | 23.1 | 34.4
  FUM6 (>=6 pt increase): number analyzed (Participants) | 88 | 119
  FUM6 (>=6 pt increase) | 29.5 | 43.7
  FUM12 (>=6 pt increase): number analyzed (Participants) | 61 | 100
  FUM12 (>=6 pt increase) | 26.2 | 47.0
  FUM18 (>=6 pt increase): number analyzed (Participants) | 45 | 83
  FUM18 (>=6 pt increase) | 28.9 | 51.8
  FUM24 (>=6 pt increase): number analyzed (Participants) | 34 | 75
  FUM24 (>=6 pt increase) | 26.5 | 48.0
  Ext FUM6 (>=6 pt increase): number analyzed (Participants) | 25 | 65
  Ext FUM6 (>=6 pt increase) | 44 | 56.9
  C5D1 (>=7 pt increase): number analyzed (Participants) | 156 | 157
  C5D1 (>=7 pt increase) | 24.4 | 28.0
  FUM6 (>=7 pt increase): number analyzed (Participants) | 88 | 119
  FUM6 (>=7 pt increase) | 34.1 | 40.3
  FUM12 (>=7 pt increase): number analyzed (Participants) | 61 | 100
  FUM12 (>=7 pt increase) | 31.1 | 45.0
  FUM18 (>=7 pt increase): number analyzed (Participants) | 45 | 83
  FUM18 (>=7 pt increase) | 31.1 | 43.4
  FUM24 (>=7 pt increase): number analyzed (Participants) | 34 | 75
  FUM24 (>=7 pt increase) | 20.6 | 42.7
  Ext FUM6 (>=7 pt increase): number analyzed (Participants) | 25 | 65
  Ext FUM6 (>=7 pt increase) | 32 | 47.7

ADVERSE EVENTS:
Time Frame: Baseline up to 8.5 years
Description: Safety population included all participants who received any amount of obinutuzumab or bendamustine therapy.
Arm/Group | Bendamustine Alone | Obinutuzumab + Bendamustine
Serious Adverse Events (participants affected / at risk) | 76/203 | 91/204
Other Adverse Events (participants affected / at risk) | 194/203 | 200/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine Alone (N=203) | Obinutuzumab + Bendamustine (N=204)
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 6 (6) | 11 (17)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 6 (6)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (2) | 2 (2)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 2 (3)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (2)
PAROXYSMAL ARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
HYDROCELE (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
NECROTISING RETINITIS (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0)
ANAL FISSURE (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 0 (0)
FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (2) | 0 (0)
MELAENA (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 2 (2)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (2)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 2 (2)
CATHETER SITE PAIN (General disorders) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 2 (2) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 3 (4)
HYPERTHERMIA (General disorders) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 1 (1)
MALAISE (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 3 (3) | 6 (7)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
GRAFT VERSUS HOST DISEASE (Immune system disorders) | 0 (0) | 1 (1)
ATYPICAL PNEUMONIA (Infections and infestations) | 1 (1) | 1 (1)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 3 (3) | 1 (1)
CAMPYLOBACTER INFECTION (Infections and infestations) | 0 (0) | 1 (1)
COXSACKIE MYOCARDITIS (Infections and infestations) | 0 (0) | 1 (1)
DEVICE RELATED SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
ENCEPHALITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
ENDOCARDITIS (Infections and infestations) | 1 (1) | 0 (0)
ERYSIPELAS (Infections and infestations) | 0 (0) | 1 (1)
ESCHERICHIA SEPSIS (Infections and infestations) | 0 (0) | 2 (2)
FUNGAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 1 (1) | 0 (0)
HEPATITIS B REACTIVATION (Infections and infestations) | 1 (1) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 3 (3) | 1 (1)
INFECTION (Infections and infestations) | 2 (2) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (5) | 3 (3)
LUNG INFECTION (Infections and infestations) | 1 (1) | 2 (2)
LUNG INFECTION PSEUDOMONAL (Infections and infestations) | 1 (2) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 2 (2) | 1 (1)
PNEUMONIA (Infections and infestations) | 12 (12) | 7 (7)
PNEUMONIA CYTOMEGALOVIRAL (Infections and infestations) | 1 (1) | 0 (0)
PSEUDOMONAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
PSEUDOMONAS BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (2)
SEPSIS (Infections and infestations) | 7 (7) | 6 (6)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1) | 2 (2)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 3 (3)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
VASCULAR DEVICE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 3 (3) | 7 (7)
JAW FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL BILE LEAK (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SEROMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
STAB WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1)
BORRELIA TEST (Investigations) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRONCHIAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CHOLANGIOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
INTESTINAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LEIOMYOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
POLYCYTHAEMIA VERA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
T-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
AMYOTROPHIC LATERAL SCLEROSIS (Nervous system disorders) | 0 (0) | 1 (1)
CENTRAL NERVOUS SYSTEM LESION (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 2 (2) | 0 (0)
POST HERPETIC NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 2 (2)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
MANIA (Psychiatric disorders) | 0 (0) | 1 (1)
DYSURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
END STAGE RENAL DISEASE (Renal and urinary disorders) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CHYLOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
PARANEOPLASTIC PEMPHIGUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SOCIAL PROBLEM (Social circumstances) | 1 (1) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine Alone (N=203) | Obinutuzumab + Bendamustine (N=204)
ANAEMIA (Blood and lymphatic system disorders) | 34 (41) | 23 (36)
NEUTROPENIA (Blood and lymphatic system disorders) | 59 (103) | 74 (150)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 50 (101) | 26 (54)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 11 (12) | 6 (6)
ABDOMINAL PAIN (Gastrointestinal disorders) | 20 (23) | 16 (18)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 15 (19) | 11 (12)
CONSTIPATION (Gastrointestinal disorders) | 40 (55) | 42 (56)
DIARRHOEA (Gastrointestinal disorders) | 61 (83) | 57 (81)
DRY MOUTH (Gastrointestinal disorders) | 12 (15) | 8 (8)
DYSPEPSIA (Gastrointestinal disorders) | 9 (11) | 13 (16)
NAUSEA (Gastrointestinal disorders) | 123 (227) | 107 (210)
VOMITING (Gastrointestinal disorders) | 54 (87) | 44 (67)
ASTHENIA (General disorders) | 25 (35) | 31 (44)
CHEST PAIN (General disorders) | 4 (4) | 11 (11)
CHILLS (General disorders) | 21 (24) | 28 (30)
FATIGUE (General disorders) | 67 (114) | 81 (151)
INFLUENZA LIKE ILLNESS (General disorders) | 9 (10) | 11 (12)
MUCOSAL INFLAMMATION (General disorders) | 8 (11) | 11 (12)
OEDEMA PERIPHERAL (General disorders) | 14 (17) | 15 (16)
PYREXIA (General disorders) | 36 (44) | 54 (80)
BRONCHITIS (Infections and infestations) | 18 (23) | 24 (36)
HERPES ZOSTER (Infections and infestations) | 14 (16) | 10 (10)
NASOPHARYNGITIS (Infections and infestations) | 8 (10) | 22 (27)
RHINITIS (Infections and infestations) | 8 (9) | 12 (13)
SINUSITIS (Infections and infestations) | 11 (14) | 24 (35)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 17 (21) | 26 (34)
URINARY TRACT INFECTION (Infections and infestations) | 12 (14) | 23 (36)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 115 (242) | 125 (283)
WEIGHT DECREASED (Investigations) | 18 (18) | 11 (11)
DECREASED APPETITE (Metabolism and nutrition disorders) | 37 (49) | 37 (40)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 15 (21) | 15 (22)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 11 (12) | 24 (31)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 18 (22) | 17 (19)
MYALGIA (Musculoskeletal and connective tissue disorders) | 15 (17) | 13 (14)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 10 (13) | 22 (27)
DIZZINESS (Nervous system disorders) | 17 (23) | 14 (22)
DYSGEUSIA (Nervous system disorders) | 16 (20) | 15 (20)
HEADACHE (Nervous system disorders) | 32 (37) | 27 (36)
INSOMNIA (Psychiatric disorders) | 21 (26) | 21 (24)
COUGH (Respiratory, thoracic and mediastinal disorders) | 40 (46) | 64 (85)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 23 (28) | 26 (27)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 17 (18)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 12 (15)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 11 (11)
PRURITUS (Skin and subcutaneous tissue disorders) | 12 (13) | 29 (38)
RASH (Skin and subcutaneous tissue disorders) | 24 (27) | 28 (35)
HYPOTENSION (Vascular disorders) | 1 (2) | 23 (26)
PHLEBITIS (Vascular disorders) | 13 (14) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.